CLINICAL TRIAL: NCT05935709
Title: Disease Stratification in GCA and PMR to Inform Management and Reduce Disease and Treatment-related Damage
Brief Title: DANIsh VASculitis Database (DANIVAS)
Acronym: DANIVAS
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Regionshospitalet Horsens (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Holbaek Sygehus (Other); Rigshospitalet, Denmark (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: DANIVAS
Record Dates: First submitted 2023-06-01; First posted 2023-07-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-04

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatica
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this national pragmatic observational study is to investigate whether the use of new diagnostic imaging modalities facilitates disease stratification that can potentially predict treatment response, relapse risk and complications and hence guide management strategies to improve disease control and reduce disease and treatment related damage.

DETAILED DESCRIPTION:
BACKGROUND Giant cell arteritis (GCA) is the most common vasculitis of the elderly. The concomitant disease polymyalgia rheumatica (PMR) is characterised by pain of the proximal muscles, general symptoms, and raised inflammatory markers. Only limited research has previously been performed nationally and internationally in GCA and PMR. To explore clinical practice, biomarkers, disease subsets, comorbidities, and long-term effectiveness of new treatments the establishment of large registries are highly warranted.

OBJECTIVES Primary objective: To compare cumulative GC doses in patients with c-GCA as compared to Large vessel (LV) -GCA

Key secondary objectives:

1. To compare cumulative GC doses in patients with pure PMR compared to PMR patients with subclinical LV-GCA
2. To compare the incidence of aortic dilatation 2 years after diagnosis in patients with c-GCA as compared to LV-GCA
3. In the subpopulation of patients whom a diagnostic Fluor-Deoxy-Glucose Positron Emissions Tomography ( FDG- PET)/CT was performed, to evaluate the risk of aortic complications (aneurisms and dissections) in GCA patients with aortic involvement as compared to patients without aortic involvement.

Once the database is established nationally, the database will be the basis for additional research projects in the future.

METHODS Using RedCap database infrastructure, clinical data including imaging will be documented in the individual Case Report Form developed by the project steering group.

The study population can be enrolled at any point during disease course and registered as either incidents ( up until 3 months from diagnosis) or prevalent. The treatment and follow up will be performed according to the National Danish GCA and PMR guidelines. At some of the visits data entry to the database will be performed: Enrollment visit, response visit(after 2 months), routine visit(after 6 months for incident patients and every year following), screening visit(2 years after diagnosis) and withdrawal visits. The aim is to include all rheumatic departments in Denmark.

Data audit to secure a high completeness will be performed regularly by a project manager the first two years and thereafter by a datamanager. Linkage of data across nationwide medical and administrative registries at the individual level will be performed. Blood samples will be collected by the infrastructure of the clinical biobank Danish ReumaBiobank (DRB).

ELIGIBILITY:
Inclusion Criteria:

* Are diagnosed with GCA or PMR within the last 5 years
* Diagnosis is established by or confirmed by a rheumatologist (clinical expert opinion)
* Speak and understand Danish
* Are able to give signed and dated informed consent

Exclusion Criteria:

* Denies or are not able to give informed consent
* Are diagnosed with other systemic autoimmune diseases that out-rules the diagnosis of GCA or PMR

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients can be included at any time during the disease course. Patients will be registered as either incident (newly diagnosed within the last 3 months) or prevalent (included during routine follow-up > 3 months after diagnosis) cases.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2051-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative glucocorticoid doses compared between patients with cranial GCA and patients with Large Vessel-GCA | From date of diagnosis with GCA until one year after. Assessed yearly up to 120 months
  based on redeemed prescriptions

SECONDARY OUTCOMES:
Comparison of cumulative glucocorticoid doses in patients with pure PMR compared to PMR with subclinical LV-GCA | From date of diagnosis with PMR until one year after. Assessed yearly up to 120 months
  based on redeemed prescriptions
Incidence of aortic dilatation in patients with c-GCA as compared to LV-GCA | 2 years after diagnosis
  Aortic dilatation is defined as diameters above the 90th percentile of the respective aortic region.The angiography can be performed as either CT or MR angiography and will be performed according to local set-up and imaging acquisition protocols.
Risk of aortic complications (aneurisms and dissections) in GCA patients with aortic involvement as compared to patients without aortic involvement. | 2 years after diagnosis
  The PET/CT scan at diagnosis compared to scan at year 2

CONTACTS AND LOCATIONS:
Overall Officials: Berit Dalsgaard Nielsen, Ass prof, Principal Investigator — Led og Bindevæv, Aarhus University Hospital, Palle Juul-Jensens Boulevard 59, 8200 Aarhus N, DK
Locations (2):
- Denmark (2):
  - Led og Bindevævssygdomme, Aarhus University Hospital, Aarhus
  - Medicinsk klinik 2, Regionshospitalet Horsens, Horsens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen BD, Kristensen S, Donskov A, Terslev L, Dreyer LW, Colic A, Hetland ML, Hojgaard P, Ellingsen T, Hauge EM, Chrysidis S, Keller KK. The DANIsh VASculitis cohort study: protocol for a national multicenter prospective study including incident and prevalent patients with giant cell arteritis and polymyalgia rheumatica. Front Med (Lausanne). 2024 Jul 3;11:1415076. doi: 10.3389/fmed.2024.1415076. eCollection 2024. PMID 39026552